CLINICAL TRIAL: NCT06137729
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of PF-07899895 Administered as Immediate and Modified Release Formulations in Healthy Adult Participants
Brief Title: A Study to Learn How the Study Medicine PF-07899895 Are Tolerated and Act in the Body of Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated early . This decision was not due to any safety concerns associated with PF-07899895 but rather due to a business decision.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C5471001; 2023-507354-32-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07899895 (Experimental): Participants will receive single or multiple ascending oral doses of PF-07899895.
  Interventions: Drug: PF-07899895
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07899895 — Participants will receive oral ascending doses.
  Arms: PF-07899895
Drug: Placebo — Participants will receive matching placebo.
  Arms: Placebo

SUMMARY:
The purposes of the study are as follows:

* To understand how safe and tolerable are different amounts of study medicine (PF-07899895).
* To measure the amount of PF-07899895 in blood after the medicine is taken by mouth.

The study is seeking participants who:

* Are male or female of 18 to 65 years of age.
* Are in good health condition.
* Have not had viral infections (HIV, HBV, or HCV). HIV, human immunodeficiency virus. - HBV, human hepatitis B virus. HCV, human hepatitis C virus.
* Have tested negative for tuberculosis.

Participants will receive either PF-07899895 or placebo (dummy pill) by chance. In the first part of the study (Part A):

* each participant will receive a total of up to 5 doses of the medicine or placebo with at least 5 days between each dose.
* after each dose, participants will stay in study clinic for 3 to5 days.

In the second part of the study (Part B):

- each participant will need to take 10 days of dosing and will stay in the study clinic for clinical checks for 13 days.

In the third part of the study (Part C):

* In SD cohort, each participant will receive a total of up to 5 doses of the medicine or placebo with at least 7 days between each dose. After each dose, participants will stay in study clinic for 5 days.
* In MD cohorts, each participant will need to take 10 days of dosing and will stay in the study clinic for clinical checks for 13 days.

The planned duration of participation from screening to follow-up in:

* Part A of the study is up to 15 to 18 weeks.
* Part B of the study is up to 11 weeks.
* Part C of the study is up to 15 to 18 weeks. Participants will also have their blood collected by the study doctors for several times.

ELIGIBILITY:
Inclusion Criteria:

* Participants, male or female, must be 18 to 65 years of age, inclusive, at the time of signing the ICD.
* BMI of 16 to 32 kg/m2; and a total body weight>50 kg (110 lb).
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs assessments, oral temperature, 12-lead ECGs, and laboratory tests.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, bowel resection) or gastrointestinal (GI) transit time (eg, constipation).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb); positive or indeterminate QuantiFERON test for tuberculosis. Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of undesired reactions to the sun (photosensitivity).
* Recent exposure to live or attenuated vaccines within 28 days of the screening visit.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention, with the exception of moderate or strong cytochrome P450 3A (CYP3A) inducers or inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of PF-07899895 used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
AE observed after single or multiple doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
  number of participants experience AE or SAEs.
Laboratory abnormalities following single or multiple ascending doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
  number of participants with laboratory abnormalities
Vital sign changes following single or multiple ascending doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
  Number of participants with change from baseline in vital signs
ECG changes following single or multiple ascending doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
  Number of participants with change from baseline in electrocardiogram (ECG) parameters
Changes in physical examination after single or multiple ascending doses | Day 1 up to Day 28 (Part A)/Day 1 up to Day 38 (Part B)
  Number of participants with change from baseline in physical examinations (PE)

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) | Day 1 up to Day 3 (Part A)
  descriptive summary of AUClast by treatment
Dose normalized AUClast divided by dose (AUClast(dn)) | Day 1 up to Day 3 (Part A)
  descriptive summary of AUClast by treatment
Maximum Observed Plasma Concentration (Cmax) | Day 1 (Part A)/Day 1 and Day 10 (Part B)
  descriptive summary of Cmax by treatment
Dose normalized Cmax divided by dose (Cmax(dn)) | Day 1 (Part A)/Day 1 and Day 10 (Part B)
  descriptive summary of Cmax,dn by treatment
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1 (Part A)/Day 1 and Day 10 (Part B)
  descriptive summary of Tmax by treatment
Area under the concentration time-profile from time 0 extrapolated to infinity (AUCinf) | Day 1 up to Day 3 (Part A)
  descriptive summary of AUCinf by treatment
Dose normalized AUCinf divided by dose (AUCinf(dn)) | Day 1 up to Day 3 (Part A)
  descriptive summary of AUCinf,dn by treatment
Plasma elimination half-life is the time measured for the plasma concentration to decrease by one half (t½) | Day 1 up to Day 3 (Part A)/Day 10 up to Day 12 (Part B)
  descriptive summary of t1/2 by treatment
Apparent clearance (CL/F) | Day 1 up to Day 3 (Part A)/Day 10 up to Day 12 (Part B)
  descriptive summary of CL/F by treatment
Apparent volume of distribution after oral dose is influenced by the fraction absorbed (Vz/F) | Day 1 up to Day 3 (Part A)/Day 10 up to Day 12 (Part B)
  descriptive summary of Vz/F
Area under the concentration-time curve from time 0 to time tau, where tau=24 hrs (AUCtau) | Day 1 and Day 12 (Part B)
  descriptive summary of AUCtau
Dose normalized AUCtau divided by dose (AUCtau(dn)) | Day 1 and Day 12 (Part B)
  descriptive summary of AUCtau,dn
Observed accumulation ratio for Rac for AUC | Day 1 and Day 12 (Part B)
  descriptive summary of observed Rac for AUC
Observed accumulation ratio for Cmax (Rac,Cmax) | Day 1 and Day 12 (Part B)
  descriptive summary of Rac,Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5471001